CLINICAL TRIAL: NCT05407948
Title: The Interaction Between Cognitive Reserve and Neuropsychological Variables, Variables Related to Psychological Well-being and Health Care Usage in Relation to Long-term Outcome After Stroke or Traumatic Brain Injury
Brief Title: The Effect of Cognitive Reserve on Outcome After Stroke or Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Natascha Ekdahl (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Natascha Ekdahl, Principal investigator, Region Gävleborg
Organization: Region Gävleborg (Other)
Other Study IDs: NESandvikenstudy
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Traumatic Brain Injury; Stroke
Keywords: Neuropsychology; Cognitive reserve; Return-to-work
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A long-term follow-up study of patients who acquired a stroke or traumatic brain injury (TBI) 5-15 years ago.

Primary objective is to describe the interaction between measures of cognitive reserve and neuropsychological variables, psychological variables and healthcare usage in relation to outcome (i.e work return, satisfaction with life, psychological well-being and overall outcome) after stroke or traumatic brain injury.

Secondary objectives are to describe differences in fatigue related to cognitive reserve after stroke or TBI and to describe differences in health-care usage related to cognitive reserve after stroke or TBI.

DETAILED DESCRIPTION:
Stroke and traumatic brain injury (TBI) are the most common causes of acquired brain injury, affecting 30000 and 25000 persons in Sweden per year respectively. According to a review article approximately 50 % of patients does not return to work after their stroke and even among patients with the least severe form of TBI, mild TBI, 10-45 % report long-term impairments. This is an indication that a considerable proportion of patients with stroke or TBI does not make a full recovery and live for many years with cognitive, physical and/or emotional impairments.

Earlier studies have found that long-term outcome after both TBI and stroke are determined by a complex combination of injury-related, demographic and neuropsychological factors. This combination is complex enough to avoid revelation of any multivariable prognostic model that can adequately predict patient outcome, despite considerable efforts. Further studies are therefore needed to improve the currently unsatisfactory possibilities of identifying patients at risk of poor outcome.

Previous research suggests that one of the reasons why people suffer differently from what appear to be similar brain injuries has to do with cognitive ability before injury, the so-called cognitive reserve. According to the theory of cognitive reserve, a high premorbid level functions as a cognitive reserve and this leads to the brain network having greater resistance to damage The protective effect of cognitive reserve is seen in many neurological conditions e.g. Alzheimer's. Common measures of cognitive reserve is education level before injury or measures of crystallized intelligence, i.e. knowledge gained through prior learning, by for instance tests of vocabulary.

Cognitive reserve as measured by education had been linked to various differences in outcome after TBI and stroke, for instance: lower education is also associated with lower probability of returning to work after both TBI and stroke, higher education is linked to higher life satisfaction and less depression. Cognitive reserve is also strongly linked to results on neuropsychological test which in turn also seem to be related to outcome after brain injury. At a group level, lower performance on cognitive tests indicates a lower probability of returning to work after injury although this is not a consistent finding. Given that education both seem to impact the susceptibility of the brain to injury and results on neuropsychological tests it is important to take education into consideration when studying the relationship between outcome on neuropsychological tests and return to work after brain injury. In previous studies it is common to control for educational level when investigating the relationship between return to work and results on neuropsychological tests but to our knowledge no-one has looked at whether neuropsychological variables have different significance för work return in different groups based on level of education.

As cognitive reserve is not only related to result on cognitive tests but also to psychological well-being, it would be of interest to investigate whether cognitive reserve interacts with measures of psychological well-being over time and how this is related to more functional measures of outcome after stroke and TBI.

Furthermore higher educational level has been found to be strongly related to better health overall but also to higher health care consumption. This apparent contradiction can in part be explained by higher usage of preventive health care services and more use of specialized health care compared to general practitioners among people with higher levels of education. For brain injury, focus of studies of health care usage have frequently been the relationship between health care usage and insurance compensation processes. A better understanding of how cognitive reserve influences health service utilization after brain injury, and how this is related to outcome, could be of value in ensuring more equal access to brain injury rehabilitation.

The aim of the current study is to examine the interaction of cognitive reserve with neuropsychological measures, variables related to psychological well-being and variables related to health care usage on long-term outcome after acquired brain injury (TBI or stroke). The study also aims to investigate whether there are differences in health-care consumption and levels of fatigue based on educational level after stroke or TBI.

STUDY SETTING The Brain Injury Rehabilitation Team in Sandviken is a specialized outpatient rehabilitation team for patients of working age with an acquired brain injury in Region Gävleborg. Interviews with the participants was conducted by telephone.

PATIENT CHARACTERISTICS Former patients at the Brain Injury Rehabilitation Team in Sandviken, Sweden, who had suffered a stroke or a traumatic brain injury between the years 2003-2016 were invited to participate in the study. The study was approved by the Regionala Etikprövningsnämnden Uppsala (2018/242, 2020-05887, 2021-02002). All participants provided written informed consent.

SAMPLE SIZE Multiple linear and logistic regression will be used in the statistical analysis. In order to achieve 80 % power, with a significance level set at p<.05 and 3 prognostic variables, 76 participants are needed to discern medium effects.

RECRUITMENT In total 236 patients fulfilled the inclusion criteria and were asked by mail if they wished to participate in the study. Of these 87 accepted and was booked for a telephone interview but only 83 were interviewed, as the remaining 4 was unreachable, in spite of repeated efforts. Chart review of the recruited participants showed that 2 of the recruited participants had an intellectual disability and one had suffered from a new brain injury. These 3 participants were therefore excluded.

DATA COLLECTION AND MANAGEMENT After receiving written consent a structured telephone interview were booked with the patient. The interview followed a standardized manual including questions about employment, overall outcome was assessed with Glasgow Outcome Scale - Extended (GOSE) life satisfaction according to Life Satisfaction Questionnaire (LiSat-11), anxiety and depression according to Hospital and Anxiety Scale (HADS). The interview was approximately 30 minutes and was carried out by a social worker, psychologist or a psychology student with no previous relation to the patient. Information concerning profession, education and level of consciousness according to Glasgow Coma Scale (GCS) or Reaction Level Scale (RLS) at the time of injury where collected from patient charts. Neuropsychological variables (including working memory index, processing speed index, Vocabulary score, Information score, Block Design score, Matrices score and Similarities score from the Wechsler scales) along with results on HADS and LiSat-11 at the time of admittance to the Brain Injury Team were also collected from patient charts through retrospective chart review. Data of health service utilization, containing information about number of visits, year and clinic, were collected from the administrative records of Region Gävleborg. Data of health service utilization were collected from three years before injury until four years after injury.

MEASURES GLASGOW OUTCOME SCALE-EXTENDED (GOSE) Glasgow Outcome Scale Extended is a global assessment of functioning after acquired brain injury. It is considered the measure of choice in TBI but is also commonly used after stroke and covers areas of independence, work, social, and leisure activities, and participation in social life. The scale consists of an 8-point ordinal scale divided into upper and lower levels of good recovery (7, 8), moderate disability (5, 6), severe disability (3, 4), vegetative state (2), and death (1).

LIFE SATISFACTION QUESTIONNAIRE (LISAT-11) Life Satisfaction Questionnaire (LiSat-11) consists of 11 questions. The instrument assesses overall satisfaction with life with one question as well as domain-specific satisfaction within ten domains, for instance mental health, ability to manage oneself, finances, with one question each. The response options extend over six levels from "Very unsatisfactory" to "Very satisfactory". LiSat-11 has been found to be valid for the general population as well as for people with acquired brain injury. The answers can be dichotomized into two groups, satisfied (options 5 and 6) and unsatisfied (options 1 to 4).

HOSPITAL ANXIETY AND DEPRESSION SCALE (HADS) The Hospital Anxiety and Depression Scale (HADS) comprises of two separate scales for anxiety and depression. Scores range from 0 to 21, with scores from 0 to 7 representing a "normal," 8-10 a "mild," 11-14 a "moderate," and 15-21 a "severe" level of anxiety or depression. The HADS has been widely used to assess anxiety and depression following TBI.

WECHSLER SCALES The Wechsler Adult Intelligence scale (WAIS) and Wechsler Memory Scale (WMS) are well-known instruments for measuring cognitive function. Both WAIS and WMS are translated and standardized för a Swedish population, In WAIS you can calculate a full scale IQ-score as well as four different indices, verbal understanding, perceptual organization, speed and working memory. In WMS-III eight primary memory indices can be calculated, one of which is a working memory index, comparable with the working memory index in WAIS. Speed index has been shown to be especially sensitive to brain damage. Also on working memory index, people with brain damage generally perform worse than controls. The individual tests subtests Vocabulary and Information seem less sensitive to brain damage and have in previous studies been used as measures of pre-morbid IQ.

DATA MANAGEMENT All data material will be recorded with a participant ID and will be unidentifiable. Only the first author will have access to the list that link participant ID with names. De-identified data will be electronically stored on the server at Region Gävleborg and will be deleted 5 years after the project has ended. The final dataset will be available to researchers actively contributing to statistical analyses and publications. Data entry will be controlled by initial exploratory analyses, including range checks, in order to promote data quality.

CONFIDENTIALTY Information on participants will be handled by health care professionals adhering to Swedish Law ensuring confidentiality and data protection. Results and data will be presented at a group level in publications, rendering identification of individual patients impossible. All data will be stored in accordance with the General Data Protection Regulation (GDPR).

STATISTICAL ANALYSIS Descriptive statistics will be used to depict demographics, injury characteristics, results on neuropsychological tests and psychological screening instruments. Multiple linear and logistic regression will be used in order to detect any interaction effect between measures of cognitive reserve and neuropsychological variables, injury-related variables and variables related to psychological well-being on the outcome variables. Power analysis show that in order to achieve 80 % power, with an alpha-level of 0.05, and three controlling variables in the regression model, the regression analysis require 76 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke or TBI between the years 2003-2016
2. Previous or ongoing contact with the outpatient brain injury rehabilitation team in Region Gävleborg
3. Currently living in Region Gävleborg. -

Exclusion Criteria:

Patients with an intellectual disability (IQ>70) or who have acquired a new brain injury will be excluded -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former patients at the Brain Injury Rehabilitation Team in Sandviken, Sweden, who had suffered a stroke or a traumatic brain injury between the years 2003-2016 were invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Return to work | 5-15 years after injury
  Degree of return to work according to degree of health insurance benefit received by the Swedish Social Insurance Agency
Life Satisfaction Scale (LiSat-11) | 5-15 years after injury
  Life Satisfaction with life overall as well as with specific areas of life. Each area is grade on a scale from 1 to 6 where higher score indicates better satisfaction.

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 5-15 years after injury
  Overall outcome after brain injury on a scale from 1 to 8, where 1 is death and 8 is upper level of good recovery
Hospital Anxiety and Depression Scale (HADS) | 5-15 years after injury
  Screening of depression and anxiety, higher scores indicate more severe problems
Fatigue | 5-15 years after injury
  Fatigue graded on a 1 to 10 visual/analog-scale (VAS) by the patients themselves in combination with the Telephone interview. 1 is no fatigue and 10 is severe fatigue
Health care consumption | 3 years before injury to 4 years after injury
  Number of contacts with the Health services in Region Gävleborg gathered from administrative systems

CONTACTS AND LOCATIONS:
Locations (1):
- Sandvikens närsjukhus, Sandviken, Gävleborg County, Sweden

IPD SHARING:
Plan to Share IPD: No
In order to fulfill the requirements of the ethical approvement of the study, results and data will be presented at a group level in publications, rendering identification of individual patients impossible

REFERENCES:
- [Background] Socialstyrelsen,
- [Background] Stenberg M, Koskinen LD, Jonasson P, Levi R, Stalnacke BM. Computed tomography and clinical outcome in patients with severe traumatic brain injury. Brain Inj. 2017;31(3):351-358. doi: 10.1080/02699052.2016.1261303. Epub 2017 Feb 16. PMID 28296529
- [Background] Harris C. Return to work after stroke: a nursing state of the science. Stroke. 2014 Sep;45(9):e174-6. doi: 10.1161/STROKEAHA.114.006205. Epub 2014 Jul 10. No abstract available. PMID 25013019
- [Background] Ahman S, Saveman BI, Styrke J, Bjornstig U, Stalnacke BM. Long-term follow-up of patients with mild traumatic brain injury: a mixed-method study. J Rehabil Med. 2013 Sep;45(8):758-64. doi: 10.2340/16501977-1182. PMID 24002311
- [Background] A. Ruet et al.,
- [Background] Silverberg ND, Gardner AJ, Brubacher JR, Panenka WJ, Li JJ, Iverson GL. Systematic review of multivariable prognostic models for mild traumatic brain injury. J Neurotrauma. 2015 Apr 15;32(8):517-26. doi: 10.1089/neu.2014.3600. Epub 2015 Jan 13. PMID 25222514
- [Background] Stern Y. What is cognitive reserve? Theory and research application of the reserve concept. J Int Neuropsychol Soc. 2002 Mar;8(3):448-60. PMID 11939702
- [Background] Barulli D, Stern Y. Efficiency, capacity, compensation, maintenance, plasticity: emerging concepts in cognitive reserve. Trends Cogn Sci. 2013 Oct;17(10):502-9. doi: 10.1016/j.tics.2013.08.012. Epub 2013 Sep 7. PMID 24018144
- [Background] M. Matérne, T. Strandberg, and L. O. Lundqvist,
- [Background] Waljas M, Iverson GL, Lange RT, Liimatainen S, Hartikainen KM, Dastidar P, Soimakallio S, Ohman J. Return to work following mild traumatic brain injury. J Head Trauma Rehabil. 2014 Sep-Oct;29(5):443-50. doi: 10.1097/HTR.0000000000000002. PMID 24263178
- [Background] Oldenburg C, Lundin A, Edman G, Nygren-de Boussard C, Bartfai A. Cognitive reserve and persistent post-concussion symptoms--A prospective mild traumatic brain injury (mTBI) cohort study. Brain Inj. 2016;30(2):146-55. doi: 10.3109/02699052.2015.1089598. Epub 2015 Nov 30. PMID 26618716
- [Background] M. D. Lezak, D. B. Howieson, D. W. Loring, J. H. Hannay, and J. S. Fischer,
- [Background] Spitz G, Ponsford JL, Rudzki D, Maller JJ. Association between cognitive performance and functional outcome following traumatic brain injury: a longitudinal multilevel examination. Neuropsychology. 2012 Sep;26(5):604-12. doi: 10.1037/a0029239. Epub 2012 Jul 16. PMID 22799747
- [Background] Stenberg M, Godbolt AK, Nygren De Boussard C, Levi R, Stalnacke BM. Cognitive Impairment after Severe Traumatic Brain Injury, Clinical Course and Impact on Outcome: A Swedish-Icelandic Study. Behav Neurol. 2015;2015:680308. doi: 10.1155/2015/680308. Epub 2015 Dec 9. PMID 26783381
- [Background] Davis LC, Sherer M, Sander AM, Bogner JA, Corrigan JD, Dijkers MP, Hanks RA, Bergquist TF, Seel RT. Preinjury predictors of life satisfaction at 1 year after traumatic brain injury. Arch Phys Med Rehabil. 2012 Aug;93(8):1324-30. doi: 10.1016/j.apmr.2012.02.036. PMID 22840830
- [Background] Rosenich E, Hordacre B, Paquet C, Koblar SA, Hillier SL. Cognitive Reserve as an Emerging Concept in Stroke Recovery. Neurorehabil Neural Repair. 2020 Mar;34(3):187-199. doi: 10.1177/1545968320907071. Epub 2020 Feb 24. PMID 32089097
- [Background] Sortso C, Lauridsen J, Emneus M, Green A, Jensen PB. Socioeconomic inequality of diabetes patients' health care utilization in Denmark. Health Econ Rev. 2017 Dec;7(1):21. doi: 10.1186/s13561-017-0155-5. Epub 2017 May 26. PMID 28550486
- [Background] Terraneo M. Inequities in health care utilization by people aged 50+: evidence from 12 European countries. Soc Sci Med. 2015 Feb;126:154-63. doi: 10.1016/j.socscimed.2014.12.028. Epub 2014 Dec 24. PMID 25562311
- [Background] Conti G, Heckman J, Urzua S. THE EDUCATION-HEALTH GRADIENT. Am Econ Rev. 2010 May;100(2):234-238. doi: 10.1257/aer.100.2.234. PMID 24741117
- [Background] Stirbu I, Kunst AE, Mielck A, Mackenbach JP. Inequalities in utilisation of general practitioner and specialist services in 9 European countries. BMC Health Serv Res. 2011 Oct 31;11:288. doi: 10.1186/1472-6963-11-288. PMID 22040155
- [Background] Kristman VL, Cote P, Yang X, Hogg-Johnson S, Vidmar M, Rezai M. Health care utilization of workers' compensation claimants associated with mild traumatic brain injury: a historical population-based cohort study of workers injured in 1997-1998. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S295-302. doi: 10.1016/j.apmr.2013.08.296. PMID 24581915
- [Background] Elbers NA, Cuijpers P, Akkermans AJ, Collie A, Ruseckaite R, Bruinvels DJ. Do claim factors predict health care utilization after transport accidents? Accid Anal Prev. 2013 Apr;53:121-6. doi: 10.1016/j.aap.2013.01.007. Epub 2013 Jan 24. PMID 23411157
- [Background] McMillan T, Wilson L, Ponsford J, Levin H, Teasdale G, Bond M. The Glasgow Outcome Scale - 40 years of application and refinement. Nat Rev Neurol. 2016 Aug;12(8):477-85. doi: 10.1038/nrneurol.2016.89. Epub 2016 Jul 15. PMID 27418377
- [Background] Fugl-Meyer AR, Melin R, Fugl-Meyer KS. Life satisfaction in 18- to 64-year-old Swedes: in relation to gender, age, partner and immigrant status. J Rehabil Med. 2002 Sep;34(5):239-46. doi: 10.1080/165019702760279242. PMID 12392240
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Teasdale G, Maas A, Lecky F, Manley G, Stocchetti N, Murray G. The Glasgow Coma Scale at 40 years: standing the test of time. Lancet Neurol. 2014 Aug;13(8):844-54. doi: 10.1016/S1474-4422(14)70120-6. PMID 25030516
- [Background] Starmark JE, Stalhammar D, Holmgren E. The Reaction Level Scale (RLS85). Manual and guidelines. Acta Neurochir (Wien). 1988;91(1-2):12-20. doi: 10.1007/BF01400521. PMID 3394542
- [Background] D. Wechsler, Wechsler Adult Intelligence Scale-III/Wechsler Memory Scale - Third Edition Technical Manual. San Antonio, TX: The Psychological Corporation, 1997
- [Background] Wilde EA, Whiteneck GG, Bogner J, Bushnik T, Cifu DX, Dikmen S, French L, Giacino JT, Hart T, Malec JF, Millis SR, Novack TA, Sherer M, Tulsky DS, Vanderploeg RD, von Steinbuechel N. Recommendations for the use of common outcome measures in traumatic brain injury research. Arch Phys Med Rehabil. 2010 Nov;91(11):1650-1660.e17. doi: 10.1016/j.apmr.2010.06.033. PMID 21044708
- [Background] Melin R, Fugl-Meyer KS, Fugl-Meyer AR. Life satisfaction in 18- to 64-year-old Swedes: in relation to education, employment situation, health and physical activity. J Rehabil Med. 2003 Mar;35(2):84-90. doi: 10.1080/16501970306119. PMID 12691338
- [Background] E. Ekstrand, J. Lexell, and C. Brogårdh,
- [Background] Hellstrom T, Kaufmann T, Andelic N, Soberg HL, Sigurdardottir S, Helseth E, Andreassen OA, Westlye LT. Predicting Outcome 12 Months after Mild Traumatic Brain Injury in Patients Admitted to a Neurosurgery Service. Front Neurol. 2017 Apr 10;8:125. doi: 10.3389/fneur.2017.00125. eCollection 2017. PMID 28443058
- [Background] van der Heijden P, Donders J. WAIS-III factor index score patterns after traumatic brain injury. Assessment. 2003 Jun;10(2):115-22. doi: 10.1177/1073191103010002001. PMID 12801182
- [Background] Carlozzi NE, Kirsch NL, Kisala PA, Tulsky DS. An examination of the Wechsler Adult Intelligence Scales, Fourth Edition (WAIS-IV) in individuals with complicated mild, moderate and Severe traumatic brain injury (TBI). Clin Neuropsychol. 2015;29(1):21-37. doi: 10.1080/13854046.2015.1005677. Epub 2015 Feb 3. PMID 25646823
- [Background] Stenberg J, Haberg AK, Follestad T, Olsen A, Iverson GL, Terry DP, Karlsen RH, Saksvik SB, Karaliute M, Ek JAN, Skandsen T, Vik A. Cognitive Reserve Moderates Cognitive Outcome After Mild Traumatic Brain Injury. Arch Phys Med Rehabil. 2020 Jan;101(1):72-80. doi: 10.1016/j.apmr.2019.08.477. Epub 2019 Sep 25. PMID 31562876
- [Background] Elkana O, Soffer S, Eisikovits OR, Oren N, Bezalel V, Ash EL. WAIS Information Subtest as an indicator of crystallized cognitive abilities and brain reserve among highly educated older adults: A three-year longitudinal study. Appl Neuropsychol Adult. 2020 Nov-Dec;27(6):525-531. doi: 10.1080/23279095.2019.1575219. Epub 2019 Mar 6. PMID 30838891

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05407948/Prot_SAP_000.pdf